CLINICAL TRIAL: NCT01732900
Title: The Predictive Value of a Gene Expression Signature in Cumulus Cells Indicative of Embryo Implantation.
Brief Title: Gene Expression in Cumulus Cells to Predict Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gema Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GEMA-201201
Record Dates: First submitted 2012-11-14; First posted 2012-11-26 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Infertility
Keywords: In vitro fertilization; Assisted reproduction; pregnancy outcome; cumulus cells
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphology (Active Comparator): Embryos selected for transfer will be based on morphology alone.
  Interventions: Other: Morphology
- GemART assay (Experimental): Embryos selected for transfer will be based upon morphology and GemART assay.
  Interventions: Other: GemART assay

INTERVENTIONS:
Other: Morphology — Embryos selected for transfer will be based upon morphology alone.
  Arms: Morphology
Other: GemART assay — Embryos selected for transfer will be based upon morphology and GemART assay.
  Arms: GemART assay

SUMMARY:
The purpose of this study is to determine the performance of a genetic assay, GemART, in cumulus cells predictive of embryo viability, and pregnancy success in women undergoing in vitro fertilization (IVF). Performance is defined as success rate per embryo transferred, as measured by the implantation rate of embryos transferred.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-39 years
* IVF cycle 1 or 2
* BMI <35
* Fertilization method: ICSI and/or IVF
* Day 3 or day 5 embryo transfer
* Treatment cycle intended for single or double embryo transfer
* Use own oocytes, not oocyte donor
* ≥ 3 embryos at final assessment
* Donor sperm acceptable
* Willing to comply with protocol and study procedures

Exclusion Criteria:

* Polycystic Ovarian Syndrome
* Presence of fibroid(s): >4 cm intramural or submucosal fibroids
* History of chemotherapy or radiation to the abdomen or pelvis
* Use of donor oocytes
* Use of reinseminated oocytes
* Preimplantation genetic diagnosis or preimplantation genetic screening during current IVF cycle
* Concurrent participation in another clinical study
* (Male): Surgically removed sperm
* (Male): <5 million sperm count

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Recorded at post-transfer week 4-9
  Clinical pregnancy, recorded as either positive or negative, will be determined using vaginal ultrasound during post-transfer week 4-9. Clinical Pregnancy rate for embryos selected using the GemART assay in conjunction with morphology will be compared with clinical pregnancy rate for embryos selected using morphology alone.

CONTACTS AND LOCATIONS:
Overall Officials: John Jarrett, MD, Principal Investigator — IVF Indiana
Locations (4):
- United States (4):
  - Reproductive Medicine Institute, Oak Brook, Illinois
  - IVF Indiana, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Reproductive Medicine Associates of Michigan, Troy, Michigan

REFERENCES:
- [Background] Iager AE, Kocabas AM, Otu HH, Ruppel P, Langerveld A, Schnarr P, Suarez M, Jarrett JC, Conaghan J, Rosa GJ, Fernandez E, Rawlins RG, Cibelli JB, Crosby JA. Identification of a novel gene set in human cumulus cells predictive of an oocyte's pregnancy potential. Fertil Steril. 2013 Mar 1;99(3):745-752.e6. doi: 10.1016/j.fertnstert.2012.10.041. Epub 2012 Nov 29. PMID 23200692